CLINICAL TRIAL: NCT03877172
Title: High Flow Nasal Cannula in Thoracic Surgery: a Physiologic Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Getinge Group (Other)
Responsible Party: Principal Investigator, Ricard Mellado Artigas, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2019/0049
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Thoracic Surgery; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-mask oxygen therapy (No Intervention): Oxygen delivered through a conventional face mask to keep saturation above 92%.
- High-flow nasal cannula (Active Comparator): High-flow nasal cannula delivered at 50 L/min and FiO2 adjusted to keep saturation above 92%.
  Interventions: Device: High-flow nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannula — To provide high-flow nasal cannula in the immediate postoperative period after lung resection surgery as compared to conventional face-mask therapy, in a randomized sequence, for 30 minutes.
  Other Names: Airvo 2, Fisher&Paykel.
  Arms: High-flow nasal cannula

SUMMARY:
The goal of this study is to evaluate the role that high-flow nasal cannulas (HFNC) have on respiratory drive, work of breathing and neuromuscular efficiency after lung resection surgery. The main question the investigators aim to answer is whether HFNC decrease respiratory drive by at least 15% in these patients, assessed by a special diaphragmatic electromyography (EMG) device (NAVA catheter). In order, to perform this study, the investigators will perform a physiological study in 40 patients. These patients will be assessed in the immediate postoperative period and HFNC will be compared to conventional face-mask therapy.

DETAILED DESCRIPTION:
Single centre, physiological crossover clinical trial in 40 patients in the immediate postoperative period after lung resection, equipped with a NAVA catheter to monitor diaphragm electrical activity (EAdi) and assess the effects that HFNC have on the respiratory drive and work of breathing as compared to conventional facemask oxygen therapy. Once in the postoperative care unit (PACU) and 1) after recovery from anaesthesia, 2) cardiorespiratory stable and 3) pain-free (see below), the intervention will start. The study will assess the effect of HFNC and oxygen via face mask on EAdi and diaphragm function, as measured by ultrasonography. HFNC and oxygen via face mask order will be randomized in a sequence (A-B or B-A) with the aid of a website (www.randomization.com). Each intervention will last for 30 minutes. The oxygen-inspired fraction (FiO2) will be adjusted to maintain a pulse oximetry (SpO2) between >92%. In the case of the high-flow nasal cannula, the study will be carried out with a flow of 50 L/min.

EAdi signal will be continuously monitored and its signal later exported to a laptop for further analysis. At the end of the 30-minute period, a blood sample will be obtained for gas analysis from the arterial line and the investigators will perform a diaphragm ultrasonography. Ultrasonography will consist of measurement of diaphragm thickness and thickening on the right side during quiet breathing and diaphragmatic excursion on both sides.

ELIGIBILITY:
Inclusion Criteria:

* Subjects submitted to lung resection with an expected mechanical ventilation time of more than 180 minutes.

Exclusion Criteria:

* Patient refusal to participate
* Contraindications to nasogastric tube placement (i.e. oesophageal varices)
* Patients less than 18 years old
* Pregnancy
* Neuromuscular disease
* Prior thoracic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-17 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory drive | Mean or median EAdi for both conditions (30 minutes each)
  Respiratory drive will be assessed as maximal EMG activity during each respiratory cycle (peak EAdi of the NAVA catheter)

SECONDARY OUTCOMES:
Thickening fraction of the right hemidiaphragm | An ultrasound will be performed 25 minutes after starting each study condition
  Diaphragm thickness will be assessed at end-inspiration and end-expiration and presented as percentage of change.
Diaphragmatic excursion | An ultrasound will be performed 25 minutes after starting each study condition
  Diaphragmatic excursion will be assessed on each side and measured in millimeters
Oxygenation | An arterial blood sample will be obtained at the end (30 min) of each study condition
  Arterial oxygen pressure to inspired oxygen fraction ratio (PF ratio)
Ventilation | An arterial blood sample will be obtained at the end (30 min) of each study condition
  Arterial pressure of carbon dioxide (CO2)
Dyspnea | Dyspnea presence by VAS will be assessed at the 30-minute mark of each condition (end of each condition) and will evaluate dyspnea for the whole condition (30 minutes).
  The presence of dyspnea will be assessed by a visual analog scale (VAS). This scale presents a range of discrete values from 0 to 10; with lower values indicating less symptoms and higher values indicating more symptoms. Participants will subjectively rate their own level of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Mellado Artigas, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided